CLINICAL TRIAL: NCT02803346
Title: Evaluation of Immunosuppression in Septic Shock: Biomarkers and Pharmacological Restoration (IMMUNOSEPSIS)
Acronym: IMMUNOSEPSIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50620
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Immunology of Septic Shock
Keywords: sepsis; septic shock; immunosuppression; HLA-DR; lymphopenia
MeSH Terms: conditions — Sepsis; Shock, Septic; Lymphopenia | interventions — Leukocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- septic shock patients
  Interventions: Other: Circulating blood (leukocytes)

INTERVENTIONS:
Other: Circulating blood (leukocytes) — mHLA-DR measurement (in vitro)

SUMMARY:
Septic syndromes (systemic inflammatory response associated with infection) remain a major although largely under-recognized health care problem and represent the first cause of mortality in intensive care units. While it has long been known that sepsis deeply perturbs immune homeostasis by inducing a tremendous systemic inflammatory response, novel findings indicate that sepsis indeed initiates a more complex immunologic response that varies over time, with the concomitant occurrence of both pro- and anti-inflammatory mechanisms. As a resultant, after a short pro-inflammatory phase, septic patients enter a stage of protracted immunosuppression. This is illustrated in those patients by reactivation of dormant viruses (CMV or HSV) or infections due to pathogens, including fungi, which are normally pathogenic solely in immunocompromised hosts. These alterations might be directly responsible for worsening outcome in patients who survived initial resuscitation as nearly all immune functions are deeply compromised. Both arms of immunity (innate and adaptive) are indeed markedly suppressed (including enhanced leukocyte apoptosis, lymphocyte anergy and deactivated monocyte functions). New promising therapeutic avenues are currently emerging from those recent findings such as adjunctive immunostimulation for the most immunosuppressed patients. The prerequisite for immunostimulation administration (IFNg, GM-CSF, IL-7) however relies on the investigators capacity in identifying the patients who could benefit from it, as there is no clinical sign of immune dysfunctions. The main objectives are:

1. to identify the best biomarkers for sepsis-induced immunosuppression and
2. to evaluate ex vivo whether drugs could rejuvenate immune functions.

ELIGIBILITY:
Inclusion Criteria:

* septic shock is defined by an identifiable site of infection, persisting hypotension despite fluid resuscitation requiring vasopressor therapy, and evidence of a systemic inflammatory response

Exclusion Criteria:

* age < 18
* immunosuppressive disease (HIV, cancer, primary immune deficiency)
* immunosuppressive treatment or corticoid treatment (dosage > 10mg/day or cumulative dose >700 mg equivalent prednisolone)
* aplasia as defined by number of circulating neutrophils < 500 cells / mm3
* extracorporeal circulation during the month prior ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: septic shock patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days post diagnosis

SECONDARY OUTCOMES:
occurrence of nosocomial infection | 28 days post diagnosis
decreased monocyte HLA-DR expression | day 3 post diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Bodinier M, Peronnet E, Brengel-Pesce K, Conti F, Rimmele T, Textoris J, Vedrine C, Quemeneur L, Griffiths AD, Tan LK, Venet F, Maucort-Boulch D, Monneret G; REALISM study group. Monocyte Trajectories Endotypes Are Associated With Worsening in Septic Patients. Front Immunol. 2021 Nov 29;12:795052. doi: 10.3389/fimmu.2021.795052. eCollection 2021. PMID 34912347